CLINICAL TRIAL: NCT04783220
Title: Comprehensive PaREnting ProgrAm to Enhance PREterm Infants' Health and Development: A Randomized Controlled Trial (PREPARE Trial)
Brief Title: PaREnting ProgrAm to Enhance PREterm Infants' Health and Development (PREPARE Trial)
Acronym: PREPARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBS-2020-0365
Record Dates: First submitted 2021-01-15; First posted 2021-03-05 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Behavioral Assessment of Children; Early Intervention
Keywords: Preterm infant; Parental stress; Early child development; Parenting in the neonatal intensive care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The parents of babies in this group will receive an educational and intervention program
  Interventions: Behavioral: Comprehensive structured parent intervention
- Control (No Intervention): The parents of babies in this group will receive the standard parent education and follow-up.

INTERVENTIONS:
Behavioral: Comprehensive structured parent intervention — 1. Educational sessions and coaching on infants' behavior cues
  2. Skills on motor stimulation
  3. Written instructions for play and stimulation activities at discharge
  4. Multidisciplinary follow-up
  5. Developmental tracking and advice via a mobile app
  Arms: Intervention

SUMMARY:
Preterm infants are at high risk of developmental delay or disabilities and they do benefit from early intervention programs. Many programs aiming at improving preterm infants' developmental outcome have been proposed with mixed results. In low to middle-income countries, clinically relevant and effective low cost interventions empowering parents have yet to be established.

DETAILED DESCRIPTION:
Education and intervention programs targeting parents of premature infants are lacking in low to middle income countries (LMIC) and in Arabic countries in particular. The main concept of this proposal is to develop a program in Arabic for parents of premature infants with the aim to increase their knowledge about short and long term problems of prematurity, increase their involvement in the care during their stay in the neonatal intensive care unit (NICU) and promote responsive and sensitive parenting in the NICU and after discharge. This is to empower parents and have them become active contributors to enhancing their infant's development through play activities and tracking of developmental milestones.

ELIGIBILITY:
Inclusion Criteria:

* Couplets of parents and their preterm infants admitted to the NICU, who are <35 weeks gestation at birth and who are deemed medically stable by their treating neonatologist.

Exclusion Criteria:

* Infants with significant neurologic disorder precluding meaningful interaction with the parents as determined by the neurologist
* Infants with major congenital anomalies precluding meaningful interaction with the parents as determined by the neurologist
* Infants with systemic medical and/ or surgical conditions precluding interaction with the parents, other than preterm-related intraventricular hemorrhage (IVH) and periventricular leukomalacia (PVL).
* Parental refusal to participate
* Absence of clearance from the neonatologist
* Infants planned to be transferred to another facility for their NICU care.

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Child developmental outcome | 9 months
  The developmental outcome of preterm children will be assessed using the Ages and Stages Questionnaire at 9 months of corrected age.
  The ASQ-3 covers 5 area of child development : Gross Motor, Fine Motor, Problem Solving, Personal-Social, Communication.
  Scores for each area should range between minimum 0 and maximum 60. Higher scores indicate that the child is developing properly.

SECONDARY OUTCOMES:
Physiological state- Respiratory rate | 1 year
  Physiological parameters including respiratory rate will be retrieved from the bedside monitors.
Physiological state - Oxygen saturation | 1 year
  Physiological parameters including oxygen saturation will be retrieved from the bedside monitors.
Neurobehavioral state | 1 year
  Behavioral state will be assessed by a cerified trained developmental specialist using a 7-point score that include: (i) Quiet/deep sleep, (ii) Active sleep, (iii) Awake State, (iv) drowsy, (v) quiet alert, (vi) active alert, (vii) crying
Parental Knowledge assessment | Before hospital discharge
  Parental knowledge assessment test will be administered before and after the education sessions using 10 true/false questions regarding topics addressed in the sessions.
Parental stress | 1 year
  The Arabic parenting stress index short form questionnaire will be used. The PSI-SF is a self-administered questionnaire and consists of 36 items divided into three subscales of 12 items each: parental distress, parent-child dysfunctional interaction and difficult child.
  For each subscales scores ranges should be between 12 and 60. For the total stress score , the minimum score is 36 and the maximum is 180. Higher scores mean more depressive symptoms.
Behavioral parenting activities | 1 year
  A questionnaire derived from the UNICEF MICS 6 questionnaire will be used. MICS or "MULTIPLE INDICATOR CLUSTER SURVEY" is a tool used to assess the activities of parents with their infants.
Parents perceptions | 1 year
  The Perceived Maternal Parenting Self-Efficacy questionnaire is a standardized valid and reliable instrument to assess parent's perceptions of their ability to care for their infants.
  PMP-SE is composed of 20 items divided into four subscales: care taking procedures, evoking behaviours, reading behaviours or signalling, and situational beliefs.
  Those items are formulated as statements using a five-point Likert scale. Scoring ranges from 20 to 80 where a higher score indicates a higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Lama Charafeddine, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Hamra, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MICS6 TOOLS — http://mics.unicef.org/tools
- See also: Agency for Healthcare Reserach and Quality (2018). NICU-2-HOME: Using Health IT to Support Parents of NICU Graduates Transitioning to Home (Illinois) | AHRQ National Resource Center; Health Information Technology: Best Practices Transforming Quality, S — http://healthit.ahrq.gov/ahrq-funded-projects/nicu-2-home-using-health-it-support-parents-nicu-graduates-transitioning-home